CLINICAL TRIAL: NCT02100930
Title: Anti-GD2 3F8 Monoclonal Antibody and GM-CSF for High-Risk Neuroblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-260
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2019-04

CONDITIONS: Neuroblastoma
Keywords: Anti-GD2 3F8 Monoclonal Antibody; oral isotretinoin; GM-CSF; Sargramostim; 13-260
MeSH Terms: conditions — Neuroblastoma | interventions — humanized 3F8 anti-GD2 monoclonal antibody; Granulocyte-Macrophage Colony-Stimulating Factor; Isotretinoin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- Neuroblastoma (Experimental): This is a single-arm, open label, open access study to provide the anti-GD2 murine IgG3 MoAb 3F8 combined with granulocyte-macrophage colony stimulating factor (GM-CSF) to patients with high-risk neuroblastoma (NB). This immunotherapy has shown efficacy against minimal residual disease (MRD) in such patients.
  Interventions: Biological: Anti-GD2 3F8 Monoclonal Antibody; Drug: GM-CSF (granulocyte-macrophage colony-stimulating factor); Drug: oral isotretinoin

INTERVENTIONS:
Biological: Anti-GD2 3F8 Monoclonal Antibody
Drug: GM-CSF (granulocyte-macrophage colony-stimulating factor)
Drug: oral isotretinoin

SUMMARY:
The purpose of this study is to be able to supply an experimental combination of drugs called 3F8 and GM-CSF (also called sargramostim) to patients with high-risk neuroblastoma who may benefit from treatment.

DETAILED DESCRIPTION:
This treatment uses 3F8/GM-CSF and isotretinoin for: Group 1 patients are in 1st CR/VGPR; Group 2 patients are in a ≥2nd CR/VGPR; and Group 3 patients have primary refractory NB in BM. All patients will receive 3F8/GM-CSF through 24 months.

Road Map/Schema for Group 1 (1st CR/VGPR) and Group 2 (≥2nd CR/VGPR) patients:

Cycle 1 3F8 (iv) + GM-CSF subcutaneous (sc) (1 wk) 2-4-wk interval Cycle 2 3F8 (iv) + GM-CSF (sc) (1 wk) 2-4-wk interval* - oral isotretinoin x14 days Cycle 3 3F8 (iv) + GM-CSF (sc) (1 wk) 2-4-wk interval - oral isotretinoin x14 days Cycle 4 3F8 (iv) + GM-CSF (sc) (1 wk) 6-8-wk interval - oral isotretinoin x14 days on, 14 days off, 14 days on Cycle 5 3F8 (iv) + GM-CSF (sc) (1 wk) 6-8-wk interval - oral isotretinoin x14 days on, 14 days off, 14 days on (6th cycle) Cycle 6 3F8 (iv) + GM-CSF (sc) (1 wk) 6-8-wk interval Cycle 7 3F8 (iv) + GM-CSF (sc) (1 wk) Continue with 6-8-wk intervals through 24 months from 1st dose of 3F8. * assessment of BM status by standard histology

Road Map/Schema for Group 3 patients (BM positive): The break between end of a cycle of 3F8/GM-CSF and start of next cycle is approximately 2-to-4-weeks through 4 cycles after achievement of CR in BM; subsequent breaks are ~6-8 weeks. Please see roadmap below for a patient achieving CR in BM after cycle 1. Cycle 1 3F8 (iv) + GM-CSF (sc) (1 wk) 2-4-wk interval* - BM negative Cycle 2 3F8 (iv) + GM-CSF (sc) (1 wk) 2-4-wk interval* - oral isotretinoin x14 days Cycle 3 3F8 (iv) + GM-CSF (sc) (1 wk) 2-4-wk interval - oral isotretinoin x14 days Cycle 4 3F8 (iv) + GM-CSF (sc) (1 wk) 2-4-wk interval - oral isotretinoin x14 days Cycle 5 3F8 (iv) + GM-CSF (sc) (1 wk) 6-8-wk interval - oral isotretinoin x14 days Cycle 6 3F8 (iv) + GM-CSF (sc) (1 wk) 6-8-wk interval - oral isotretinoin x14 days on, 14 days off, 14 days on (6th cycle) Cycle 7 3F8 (iv) + GM-CSF (sc) (1 wk) 6-8-wk interval Continue with 6-8-wk intervals through 24 months from 1st dose of 3F8.

* assessment of BM response by standard histology

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by international criteria,62 i.e., histopathology (confirmed by the MSKCC Department of Pathology) or BM metastases plus high urine catecholamine levels.
* High-risk NB, as defined by risk-related treatment guidelines and the International NB Staging System, i.e., stage 4 with (any age) or without (>18 months) MYCNamplification, 63 or MYCN-amplified NB other than stage 1.64,65
* Patients are in CR/VGPR or have primary refractory NB in BM - i.e., NB resistant to standard therapy, as evidenced by persistence of NB in BM by histology or MIBG scan, but all other findings in scans show VGPR.
* Children and adults are eligible.
* Signed informed consent indicating awareness of the scheduling and side effects, as well as testing requirements, of this program.

Exclusion Criteria:

* Existing severe major organ dysfunction, i.e., renal, cardiac, hepatic, neurologic, pulmonary, or gastrointestinal toxicity > or = to grade 3, except for grade 3 hematologic toxicity.
* Progressive disease (PD)
* History of allergy to mouse proteins.
* Active life-threatening infection.
* Human anti-mouse antibody (HAMA) titer >1000 Elisa units/ml.
* Pregnant women
* Inability to comply with protocol requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-03; Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Neuroblastoma: This is a single-arm, open label, open access study to provide the anti-GD2 murine IgG3 MoAb 3F8 combined with granulocyte-macrophage colony stimulating factor (GM-CSF) to patients with high-risk neuroblastoma (NB). This immunotherapy has shown efficacy against minimal residual disease (MRD) in such patients.
  Anti-GD2 3F8 Monoclonal Antibody
  GM-CSF (granulocyte-macrophage colony-stimulating factor)
  oral isotretinoin
Period: Overall Study
Arm/Group | Neuroblastoma
Started | 69
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neuroblastoma
Number analyzed (Participants) | 69
Age, Continuous [Median (Full Range); unit: years] | 4 [1 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 68
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 52
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Response
Description: Disease status is defined by the International Neuroblastoma Response Criteria - Complete response/remission (CR): NED; Partial response/remission: >50% decrease in all disease parameters, exceptbone scan unchanged or improved; no more than 1 positive bone marrow site; Stable disease: <50% decrease in all tumor markers; Progressive disease (PD): new lesion, or >25 % increase in any disease marker.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Neuroblastoma
Number analyzed (Participants) | 69
Participants
  No Evidence of Disease | 40
  Complete Response | 3
  Partial Response | 1
  Stable Disease | 6
  Progression of Disease | 19

2. Primary Outcome: Complete Remission
Description: as for outcome 1
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Neuroblastoma
Number analyzed (Participants) | 69
Participants
  No Evidence of Disease | 40
  Complete Response | 3
  Partial Response | 1
  Stable Disease | 6
  Progression of Disease | 19

ADVERSE EVENTS:
Time Frame: 2 year
Arm/Group | Neuroblastoma
All-Cause Mortality (participants affected / at risk) | 16/69
Serious Adverse Events (participants affected / at risk) | 26/69
Other Adverse Events (participants affected / at risk) | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neuroblastoma (N=69)
Abdominal Pain (Gastrointestinal disorders) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever (General disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 3
Hypothermia (General disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Infections and infestations - Other, specify (Infections and infestations) | 8
Intracranial hemorrhage (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Resp, thoracic & mediastinal disorder Other, spec (Respiratory, thoracic and mediastinal disorders) | 2
Skin infection (Infections and infestations) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
White blood cell decreased (Investigations) | 1
Wound infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neuroblastoma (N=69)
Edema face (General disorders) | 6
Pain (General disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 6
Urticaria (Skin and subcutaneous tissue disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Flushing (Vascular disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Agitation (Psychiatric disorders) | 4
Hypotension (Vascular disorders) | 4
Anxiety (Psychiatric disorders) | 3
Hypertension (Vascular disorders) | 3
Localized edema (General disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Fever (General disorders) | 2
Headache (Nervous system disorders) | 2
Irritability (Psychiatric disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Oral pain (Gastrointestinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT02100930/Prot_SAP_000.pdf